CLINICAL TRIAL: NCT02987504
Title: A Multicenter, Dose-Escalation, Phase 1 Study of Samalizumab (ALXN6000) to Evaluate the Pharmacokinetics, Safety, and Tolerability in Patients With Advanced Cancer
Brief Title: Study of Samalizumab in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN6000-ONC-102
Record Dates: First submitted 2016-11-18; First posted 2016-12-09 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Solid tumor; Phase 1
MeSH Terms: conditions — Neoplasms | interventions — samalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Samalizumab 10, 15, 20 milligrams (mg)/kilogram (kg) Dose (Experimental): Participants received escalating doses of 10, 15, and 20 mg/kg of samalizumab IV every 21 days. Enrollment at each dose level and safety assessments were completed prior to enrolling at the next dose level; intra-participant dose escalation was not allowed.
  3 participants were enrolled into a dose cohort: If 0/3 participants developed dose limiting toxicities (DLT) within Cycle 1, enrollment began at the next higher dose to a maximum of 20 mg/kg. If 1/3 participants developed a DLT, the dose cohort was expanded to include 3 new participants. If 0/3 new participants developed a DLT within Cycle 1, enrolment began at the next higher dose level. If ≥1 of 3 new participants developed a DLT within Cycle 1, dose-escalation was terminated, and the dose level 5 mg/kg below the current dose was considered the MTD. If ≥2 of 3 participants developed DLTs within Cycle 1, dose-escalation was terminated, and the dose level 5 mg/kg below the current dose was considered the MTD.
  Interventions: Drug: Samalizumab

INTERVENTIONS:
Drug: Samalizumab — Samalizumab is a humanized, anti CD200 monoclonal antibody provided as a sterile 5 mg/milliliters (mL) solution for IV administration.
  Other Names: ALXN6000

SUMMARY:
This is a multicenter, open-label, dose-escalation, Phase 1 study of intravenous (IV) samalizumab to determine its maximum tolerated dose (MTD), overall safety/tolerability, pharmacokinetic and pharmacodynamic parameters, and efficacy in participants with advanced cancer. The study was terminated for administrative reasons and not due to any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant was ≥ 18 years of age at Screening.
2. Eastern Cooperative Oncology Group performance status of 0 to 2.
3. Participant had advanced/metastatic cancer with disease progression after treatment with all available therapies known to confer clinical benefit.
4. Participant had a life expectancy of greater than 12 weeks.

Exclusion Criteria:

1. Participant had a symptomatic brain metastasis.
2. Participant had active gastrointestinal bleeding as evidenced by either hematemesis or melena.
3. Participant had acute gastrointestinal ulcers.
4. Participant had a history of any cancer other than the present condition (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 3 years.
5. Participant with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration.
6. Participant had an active infection requiring therapy.
7. Participant's serum was positive for the presence of hepatitis B surface antigen, antibodies to hepatitis C virus, or antibodies to human immunodeficiency virus 1/2.
8. Participant had significant cardiovascular impairment (history of New York Heart Association Functional Classification system Class III or IV) or a history of myocardial infarction or unstable angina within the past 6 months prior to study drug treatment.
9. The participant's most recent test values within 14 days before the date of entry met the following standards:

   * Bone marrow function: neutrophil count ≤1500/millimeter (mm)^3, hemoglobin ≤9.0 grams/deciliter, platelet count ≤100,000/mm^3.
   * Liver function: total bilirubin ≥1.5 x the upper limit of normal (ULN) based on the standard value of each institution, aspartate aminotransferase and alanine aminotransferase ≥2.5 x ULN based on the reference laboratory.
   * Renal function: serum creatinine ≥1.5 x ULN based on the reference laboratory.
10. Participant had ongoing immune-stimulated adverse events from other immunotherapies (for example, pneumonitis, thyroiditis, or hepatitis) or a history of pneumonitis.
11. Participant had received chemotherapy, targeted therapy, and/or immunotherapy within the 28 days prior to first dose of study drug, or within a Washout Period for the chemotherapy, targeted therapy, and/or immunotherapy of 5 half-lives, whichever occurred first.
12. Participant had toxicities from previous immunotherapy that had not resolved to Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Number Of Participants Experiencing DLT Graded According To CTCAE Version 4.03, Observed In The Cycle 1 In Order To Meet The Objective Of Assessment Of The MTD | Safety monitoring began at the informed consent obtained and continued up to 28 days after the last dose of samalizumab or until new anti-tumor therapy, whichever was earlier.
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Maximum Plasma Concentration After Administration Of Samalizumab | 21 days in Cycle 1
Area Under The Plasma Drug Concentration-time Curve After Administration Of Samalizumab | 21 days in Cycle 1

SECONDARY OUTCOMES:
Objective Response Rate Using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Up to 2 Years
Disease Control Rate Using RECIST 1.1 | Up to 2 Years
Duration Of Response | Up to 2 Years
Progression Free Survival | Up to 2 Years
Overall Survival | Up to last participant completing at least 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - New Haven, Connecticut
  - Grand Rapids, Michigan
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No